CLINICAL TRIAL: NCT04632511
Title: Metabotyping of Overweight and Obese Children Towards Early Detection of Insulin Resistance and Low-grade Inflammation by Means of a Rectal Sampler
Brief Title: Metabotyping of Overweight and Obese Children
Acronym: RecSAMP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: Universitaire Ziekenhuizen KU Leuven (Other); Universitair Ziekenhuis Brussel (Other); Algemeen Ziekenhuis Maria Middelares (Other); AZ Jan Palfijn Gent (Other); AZ Sint-Lucas Gent (Other); University Hospital, Antwerp (Other); AZ Alma (Other); AZ Sint-Jan AV (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: BC-06939
Record Dates: First submitted 2020-11-09; First posted 2020-11-17 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Metabolic Disease; Obesity, Infant
Keywords: metabolomics; mass spectrometry
MeSH Terms: conditions — Metabolic Diseases; Pediatric Obesity

STUDY DESIGN:
Intervention Model Description: Children with overweight and obesity and normal-weight children
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Obese group (Other): Metabolome measurements on feces and urine.
  Interventions: Device: MetaSAMP
- Children with overweight, not yet obese (Other): Metabolome measurements on feces and urine.
  Interventions: Device: MetaSAMP
- Normal-weight control group (Other): Metabolome measurements on feces and urine.
  Interventions: Device: MetaSAMP

INTERVENTIONS:
Device: MetaSAMP — Rectal Sampler

SUMMARY:
Today's children are increasingly facing metabolic-related health issues, among which the worldwide prevalence of overweight and obesity is rising at an alarming pace. Childhood obesity is associated with the early onset of chronic diseases including an emergence of prediabetes and diabetes mellitus type 2. The decline of insulin sensitivity already years before puberty, exposes children to long- term complications prior the appearance of clinical symptoms and time of diagnosis. The shortened life expectancy and large economic burden imposed underlines the need for the identification of metabotypes at risk at an early stage. One's genetics, microbial gut composition and every aspect of the environment in which children are raised have been implicated in diet-related obesity rendering metabolomics a very powerful tool towards precision medicine. Yet, the excellence of stool in reflecting the intertwining thereof is completely unexplored for pediatric purposes, whereas blood sampling causing pain and stress for child and parent only captures a narrow fraction of the metabolome. As such, rectal sampling using a customised medical swab for optimal gut metabolome coverage is envisioned. Ambient laser desorption ionisation will be hyphenated to high-resolution mass spectrometry-based metabolomics to provide a framework for elucidating predictive and/or prognostic biomarkers for ever-increasing pediatric metabolic diseases such as obesity and (pre)diabetes.

DETAILED DESCRIPTION:
The impetus for this research proposal stems from the ever-increasing metabolic-related health issues impacting today's children. Particularly, the high prevalence of childhood obesity accompanied by substantial progression to 'prediabetic state' at teen age and full-blown DMT2, the most prevailing endocrine disease worldwide, at early adulthood. Several risk factors for the development of overt DMT2 and crescent atherogenic processes, including unhealthy lifestyle patterns, decreased physical activity and (subsequent) obesity, that may be considered markers of metabolic abnormalities, such as insulin resistance, are already well-established in children with impaired glucose tolerance prior to time of diagnosis around early adolescence. Moreover, even in individuals with normal glucose tolerance, insulin resistance has been pointed out a major risk factor and predictor for the development of DMT2. Conversely, the micro- and macrovascular events do not readily appear until maturity, thereby predisposing obese children to the development of several long-term complications urging the quest for diagnostic, prognostic and/or predictive biomarkers for insulin resistance and related metabolic diseases. Hence, intervening in the pre-pubertal life stage becomes of paramount importance. As a pivotal component in precision medicine, and unlike routine measurements that only include a narrow set of blood chemistry analytes, metabolomics reveals a far more comprehensive metabolic signature. Taken together that DM and related comorbidities are considered metabolic diseases with a dysregulated lipid metabolism being a central factor in the pathogenesis, metabolomics (and in particular lipidomics) is of key importance in this research proposal. Furthermore, given the collision between genes, gut microbiota and environmental changes preceding the development of DM and, in addition, the excellence of stool in reflecting the metabolic interactions and outcomes thereof, an innovative rectal sampler using a medical swab with customized surface tip for optimal gut metabolome coverage will be used. REIMS significantly reduces time (< 10 s) and workload (minimal sample preparation), enhancing research output and efficiency. The aim is the early identification of children who are destined to develop obesity-related chronic diseases.

ELIGIBILITY:
Inclusion Criteria:

* prepubertal

Exclusion Criteria:

* no diabetes type 1 or 2, no endocrine disease, no chronic medication

COHORT NAME: MetaBEAse

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 232 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
rectal MetaSAMP | 2 years
  Fecal metabolomics vs MetaSAMP (congruence)

SECONDARY OUTCOMES:
Metabolome markers | 4 years
  predictive/prognostic value in scope of risk assessment

CONTACTS AND LOCATIONS:
Overall Officials: Jean De Schepper, Principal Investigator — University Ghent
Locations (10):
- Belgium (10):
  - Ghent University, Ghent, East-flanders
  - AZ Alma, Eeklo, Oost-Vlaanderen
  - AZ Sint-Elisabeth, Zottegem, Oost-Vlaanderen
  - OLV Lourdes Waregem, Waregem, West-Vlaanderen
  - UZA, Antwerp
  - AZ Sint-Jan Brugge, Bruges
  - General Hospital Jan-Palfijn, Ghent
  - General Hospital Sint-Lucas, Ghent
  - University Hospital Brussels, Jette
  - University Hospital Leuven, Leuven

IPD SHARING:
Plan to Share IPD: No